CLINICAL TRIAL: NCT01046994
Title: Prospective Controlled Trial on Surgical Treatment of Type 2 Diabetes Patients With BMI 25-30 by Means of Biliopancreatic Diversion
Acronym: DIA-BPD 25-30
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Santa Chiara Hospital (Other); Istituto Nazionale per lo Studio e la Cura dei Tumori (Other)
Responsible Party: Nicola Scopinaro, Professor of Surgery, Azienda Ospedaliera Universitaria San Martino
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIA-BPD
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus; Bariatric Surgery; Biliopancreatic Diversion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Biliopancreatic Diversion; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgery (Experimental): biliopancreatic diversion
  Interventions: Procedure: biliopancreatic diversion
- standard medical care (Active Comparator): patients treated according to the rules of good clinical practice
  Interventions: Drug: antidiabetics

INTERVENTIONS:
Procedure: biliopancreatic diversion — biliopancreatic diversion consists of a distal gastrectomy with a long Roux-en-Y reconstruction, where the enteroenterostomy is placed 50 cm proximal to the ileocecal valve
  Arms: surgery
Drug: antidiabetics — patients are treated with conventional antidiabetic drugs according to the rules of good clinical practice
  Arms: standard medical care

SUMMARY:
A previous prospective study of BPD effect on type 2 diabetes patients with BMI 25-35 (DIA-CHIR) showed that T2DM is less sensitive to BPD beneficial effect in the simply overweight patients. A new prospective study was then planned with the aim to gain insight in the mechanism of action of BPD in T2DM patients in the 25-30 BMI range. Thirty patients will be submitted to BPD and compared with 10 nonoperated controls. Euglycemic-hyperinsulinemic clamp, OGTT, and mixed meal test will be performed in all subjects preoperatively, and 1 month, 1 year, and 5 years after BPD. Complete clinical and biochemical evaluations will be performed at 1, 4, 8, and 12 months, and every sixth month thereafter until the end of the fifth year.

ELIGIBILITY:
Inclusion Criteria:

* age: 35-70 years
* diabetes duration: >5 years
* documented poor glycemic control (HbA1c =>8% despite medical treatment according to GCP)
* presence of comorbidities or complications (e.g. dyslipidemia, arterial hypertension, neuropathy, retinopathy, CVD, previous stroke or TIA, lower limb amputation)
* availability to comply with the entire follow-up

Exclusion Criteria:

* general contraindications to BPD (applies also to medical controls)
* presence of anti-islet or anti-GAD antibodies or plasma C-peptide concentration <0.5 mcg/L
* blindness
* severe concomitant medical conditions (e.g. liver cirrhosis, renal failure, collagen diseases, severe endocrinopathies)
* heart failure
* recent history (less than 12 months) of myocardial infarction, stroke or TIA
* unstable angina
* pregnancy
* previous or concomitant malignancy
* severe active inflammatory, neurologic, or cardiovascular conditions
* geographic inaccessibility
* any condition which, in the opinion of the Principal Investigator, may make risky the participation in the study or bias the results

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Diabetes control as defined by FSG and HbA1c | 1 year

SECONDARY OUTCOMES:
Diabetes control as defined by FSG and HbA1c | 5 years
Assessment of prevalence and severity of diabetes complications | 5 years
Assessment of patient BMI | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Martino, Genova, Italy